CLINICAL TRIAL: NCT00001232
Title: Pituitary Gonadotropin Response to GnRH Stimulation in Menstrual, Climacteric and, Menopause-Related Mood and Behavioral Disorders
Brief Title: The Effect of GnRH on Pitutitary Hormones in Menstrual-Cycle Mood Related Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 880132; 88-M-0132
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-07

CONDITIONS: Depressive Disorder; Healthy; Mental Disorders; Mood Disorders
Keywords: Depression; FSH; GnRH; LH; Menopause; Menstrual Cycle
MeSH Terms: conditions — Depressive Disorder; Mental Disorders; Mood Disorders; Depression

SUMMARY:
The normal menstrual cycle is produced by a series of hormonal signals that starts with the release of gonadotropin-releasing hormone (GnRH) from the hypothalamus. The hypothalamus is located in the brain and is often referred to as the master gland. GnRH then acts on the pituitary gland and causes it to release two hormones, follicle stimulating hormone (FSH) and lutenizng hormone (LH). LH and FSH act on the ovary and cause it to release the hormones directly involved in menstruation, estrogen and progesterone.

The purpose of this research study is to evaluate the hypothalamic-pituitary-gonadal axis activity as measured by pituitary hormones, FSH and LH in response to intravenous doses of gonadotropin releasing hormone (GnRH) in menstrual cycle-related hormones.

DETAILED DESCRIPTION:
This protocol is designed to accompany clinical protocol #81-M-0126, "The Phenomenology and Biophysiology of Menstrually Regulated Mood and Behavior Disorders", as well as the submitted protocol, "The Phenomenology and Biophysiology of Climacteric and Menopause-Related Mood and Behavioral Disorders." Its purpose will be to evaluate hypothalamic-pituitary-gonadal axis regulation as measured by pituitary gonadotropin, i.e., follicle stimulating hormone (FSH) and luteinizing hormone (LH), response to intravenous administration of gonadotropin releasing hormone (GnRH) in menstrual cycle-related mood disorders.

ELIGIBILITY:
Age 18-65.

Female.

Use of barrier methods of birth control.

Not pregnant.

Not taking ongoing medications.

No medical illnesses.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140
Dates: Start 1988-07; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rubinow DR, Hoban MC, Grover GN, Galloway DS, Roy-Byrne P, Andersen R, Merriam GR. Changes in plasma hormones across the menstrual cycle in patients with menstrually related mood disorder and in control subjects. Am J Obstet Gynecol. 1988 Jan;158(1):5-11. doi: 10.1016/0002-9378(88)90765-x. PMID 2962499
- [Background] Schmidt PJ, Gindoff PR, Baron DA, Rubinow DR. Basal and stimulated gonadotropin levels in the perimenopause. Am J Obstet Gynecol. 1996 Sep;175(3 Pt 1):643-50. doi: 10.1053/ob.1996.v175.a74255. PMID 8828428
- [Background] Fujimoto VY, Klein NA, Battaglia DE, Bremner WJ, Soules MR. The anterior pituitary response to a gonadotropin-releasing hormone challenge test in normal older reproductive-age women. Fertil Steril. 1996 Mar;65(3):539-44. PMID 8774283